CLINICAL TRIAL: NCT06520111
Title: CRISAL Study:Cancer Risk In Secreting Adrenal Lesions
Acronym: CRISAL
Status: Recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Diletta Corallino, Principal Investigator; M.D; PhD student, IRCCS San Raffaele
Other Study IDs: CRISAL (4051 CESC)
Record Dates: First submitted 2024-06-18; First posted 2024-07-25 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Adrenal Tumor; Adrenal Incidentaloma; Surgery
Keywords: cancer risk; adrenal surgery; secreting adrenal lesions
MeSH Terms: conditions — Adrenal Gland Neoplasms; Adrenal incidentaloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients underwent surgery for secreting adrenal lesion
- patients underwent surgery for non- secreting adrenal lesion

SUMMARY:
The aim of the present study is to report the cancer risk in secreting adrenal lesions. Secondary aims: to compare the incidence of cancer in secreting versus non-secreting adrenal lesions, in order to evaluate whether adrenal hormone activity can be considered an independent predictive indicator of malignancy; compare intraoperative and 30-day postoperative outcomes of patients undergoing adrenalectomy for secreting adrenal lesions versus non-secretoring lesions; regardless of the type of adrenal lesion, identify if there is one MIS adrenal approach that is superior to the others in terms of intra- and postoperative outcomes.

DETAILED DESCRIPTION:
Background: The risk of adrenal cancer increases with increasing lesion size. Up to 60% of malignant adrenal lesions have hormonal activity and that hypercortisolism is strongly suggestive of malignancy, however data regarding the risk of cancer risk in secreting adrenal lesions are not indicated.

Although guidelines suggest open adrenalectomy for lesions with preoperative features suspicious of malignancy (size ≥ 6 cm, radiological features suggestive of malignancy, history of neoplastic disease, rapid growth, several authors have reported the safety and feasibility of minimally invasive surgery (MIS) also in these cases.

Since no clear superiority of one MIS approach over another (lateral, posterior, or anterior approach) in terms of perioperative outcomes has been demonstrated, the guidelines agree on using the more familiar approach to the surgeon.

Knowing the oncological risk of adrenal secretion lesions could allow greater awareness in the patient's multidisciplinary approach and a better balance of the risk-benefit ratio in the choice of management of the patient affected by secreting adrenal lesion, especially in the case of asymptomatic lesion or manageable with medical therapy. Comparison of the various surgical approaches for the different types of adrenal lesions could allow identifying the best surgical route for each of them.

Methods: This study will be conducted in accordance with the principles of the Declaration of Helsinki and the guidelines for good clinical practice (ICH/GCP). The study protocol will be approved by the Ethics Committee of the institutions involved. An Institutional Data Safety Monitoring Board will also be appointed.This is an ambispective (retrospective and prospective) multicentre observational study. It will based on the consecutive enrollment of all patients aged 18 years or over undergoing elective adrenalectomy, after the acceptance of informed consent. For the primary aim of the study, only patients affected by secreting adrenal lesion will be considered and the incidence of cancer will be established on the basis of the definitive histology. For the further aims of the study, all enrolled patients will be divided into: patients with secreting adrenal lesions and patients with non-secreting adrenal lesions. Both groups will be stratified on the basis of definitive histology (malignant/benign) in order to identify the incidence of cancer for each group, the results will then be compared within and postoperative at 30 days. To assess the superiority of one approach over another, all patients will be stratified according to the minimally invasive approach adopted (anterior transperitoneal, lateral transperitoneal, lateral retroperitoneal, prone retroperitoneal, laparoscopic, robotic) and the type of adrenal pathology (secretory lesion, malignant tumor, metastasis, pheochromocytoma, etc…) and will be compared in terms of intra and 30 days postoperative results. All patients undergoing elective adrenalectomy aged ≥ 18 years will be included in the present study. Emergency cases and pregnant patients will be excluded.

The study involves the collection of the following data through the Redcap platform: patient demographic data, preoperative data (comorbidities and pharmacological therapies:, previous abdominal surgery, cancer history, lesion size and site, preoperative imaging and hormonal evaluation, American Society of Anaesthesiologists (ASA) class, Charlson comorbidity index (CCI) score), intraoperative data (surgical technique and surgical approach, trocar number, position and size in case of minimally invasive surgery, type of incision in case of open surgery, intraoperative complications, associated surgical procedures, conversion rate, operative time, intraoperative blood transfusions) and postoperative data (complications according to the Clavien-Dindo classification, re-intervention rate, postoperative stay, 30-day hospital readmission rate, 30 days-mortality, definitive histological examination, oncological results at follow up, participating center number of adrenalectomies by year, number of adrenalectomies per year performed by the operator.

Statistic analysis:A formal determination of the sample size was not carried out due to the ambispective observational nature of the study cohort and due to the absence in the literature of a common agreement on the incidence of cancer in patients with adrenal secreting lesions. Based on the case-series available from the SICE (Società Italiana di Chirurgia Endoscopica), a total recruitment capacity is estimated (summation of the number of patients per year per participating center), of about 300 patients.Categorical variables will be estimated as absolute and relative frequency, while continuous variables as median (IQR interquartile range). Inferential statistics for categorical variables will be estimated by Fisher exact test, while those of continuous variables by Mann-Whitney and Kruskal-Wallis tests (for independent data) and Wilcoxon and Friedman tests (for repeated data).

Institutional Review Boards. Authorship and publication: The rules described here apply to any presentation of this study. Members of the scientific committee qualify for the authorship of this study. Up to three authors per participating center can be entered into group authorship, which will be fully citable. The order of authors in the authorship group will be based on their active contribution to the study. Study results may be published and/or presented as final analyzes only after study completion. Publication and/or presentation means any paper, podium presentation, poster, abstract, or any other public presentation of this research. Data of each patient will be collected autonomously and anonymously by the single centers involved, using a common alphanumeric code decided by the coordinating centre. The collection of the aforementioned data will take place only after acceptance of the informed consent by the patient in accordance with the Declaration of Helsinki and after approval by the Ethics Committee of the proposing centre.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective adrenalectomy;
* Patients aged ≥ 18 years
* Acceptance of informed consent

Exclusion Criteria:

Patients undergoing emergency adrenalectomy;

* Patients aged ≤ 18 years
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an ambispective (retrospective and prospective) multicentre observational study. It will based on the consecutive enrollment of all patients aged 18 years or over undergoing elective adrenalectomy, after the acceptance of informed consent. For the primary aim of the study, only patients affected by secreting adrenal lesion will be considered and the incidence of cancer will be established on the basis of the definitive histology. For the further aims of the study, all enrolled patients will be divided into: patients with secreting adrenal lesions and patients with non-secreting adrenal lesions. Both groups will be stratified on the basis of definitive histology (malignant/benign) in order to identify the incidence of cancer for each group, the results will then be compared within and postoperative at 30 days.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-27 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Cancer risk in secreting adrenal lesions. | From July to December 2024
  Number of patients who underwent adrenalectomy for secreting adrenal lesion which later proved to be malignant at definitive histological examination.
  This variable will be estimated as absolute and relative frequency and percentage value

SECONDARY OUTCOMES:
Cancer risk in secreting versus non-secreting adrenal lesions | From July to December 2024
  Comparison between the incidence of cancer in patients affected by secreting adrenal lesions VS patients affected by non-secreting adrenal lesions.
  These two groups will be matched based on other preoperative characteristics (comorbidities and pharmacological therapies, cancer history, lesion size and site, preoperative imaging and hormonal evaluation) to reduce potential bias
  Categorical variables will be estimated as absolute and relative frequency, while continuous variables as median (IQR interquartile range). Inferential statistics for categorical variables will be estimated by Fisher exact test, while those of continuous variables by Mann-Whitney and Kruskal-Wallis tests (for independent data) and Wilcoxon and Friedman tests (for repeated data).
Intraoperative and postoperative outcomes of patients undergoing adrenalectomy for secreting adrenal lesions versus non-secreting lesions | From July to December 2024
  Comparison between intraoperative and 30-day postoperative outcomes of patients undergoing adrenalectomy for secreting adrenal lesions versus non-secretoring lesions.
  Categorical variables will be estimated as absolute and relative frequency, while continuous variables as median (IQR interquartile range). Inferential statistics for categorical variables will be estimated by Fisher exact test, while those of continuous variables by Mann-Whitney and Kruskal-Wallis tests (for independent data) and Wilcoxon and Friedman tests (for repeated data).
Intraoperative and postoperative outcomes in different minimally invasive adrenalectomies | From July to December 2024
  Comparison between the intraoperative and postoperative outcomes in different minimally invasive adrenalectomies (lateral, posterior, or anterior approach).
  Categorical variables will be estimated as absolute and relative frequency, while continuous variables as median (IQR interquartile range). Inferential statistics for categorical variables will be estimated by Fisher exact test, while those of continuous variables by Mann-Whitney and Kruskal-Wallis tests (for independent data) and Wilcoxon and Friedman tests (for repeated data).

CONTACTS AND LOCATIONS:
Locations (1):
- General and Mininvasive Surgery Department, Pederzoli Hospital,, Peschiera del Garda, Verona, Italy., Italy

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared among other researchers involved in the study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From January to December 2024
Access Criteria: All researchers will be involved in the IPD management through SICE (Società di chirurgia endoscopica e nuove tecnologie)
URL: https://siceitalia.com/survey-studi/studio-crisal-e-decorated/

REFERENCES:
- [Background] Fassnacht M, Johanssen S, Quinkler M, Bucsky P, Willenberg HS, Beuschlein F, Terzolo M, Mueller HH, Hahner S, Allolio B; German Adrenocortical Carcinoma Registry Group; European Network for the Study of Adrenal Tumors. Limited prognostic value of the 2004 International Union Against Cancer staging classification for adrenocortical carcinoma: proposal for a Revised TNM Classification. Cancer. 2009 Jan 15;115(2):243-50. doi: 10.1002/cncr.24030. PMID 19025987
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Birsen O, Akyuz M, Dural C, Aksoy E, Aliyev S, Mitchell J, Siperstein A, Berber E. A new risk stratification algorithm for the management of patients with adrenal incidentalomas. Surgery. 2014 Oct;156(4):959-65. doi: 10.1016/j.surg.2014.06.042. PMID 25239353
- [Background] Stefanidis D, Goldfarb M, Kercher KW, Hope WW, Richardson W, Fanelli RD; Society of Gastrointestinal and Endoscopic Surgeons. SAGES guidelines for minimally invasive treatment of adrenal pathology. Surg Endosc. 2013 Nov;27(11):3960-80. doi: 10.1007/s00464-013-3169-z. Epub 2013 Sep 10. No abstract available. PMID 24018761
- [Background] Kazaure HS, Sosa JA. Volume-outcome relationship in adrenal surgery: A review of existing literature. Best Pract Res Clin Endocrinol Metab. 2019 Oct;33(5):101296. doi: 10.1016/j.beem.2019.101296. Epub 2019 Jul 12. PMID 31331729
- [Background] undefined
- [Background] Bergamini C, Martellucci J, Tozzi F, Valeri A. Complications in laparoscopic adrenalectomy: the value of experience. Surg Endosc. 2011 Dec;25(12):3845-51. doi: 10.1007/s00464-011-1804-0. Epub 2011 Jun 17. PMID 21681621
- [Background] Kahramangil B, Kose E, Remer EM, Reynolds JP, Stein R, Rini B, Siperstein A, Berber E. A Modern Assessment of Cancer Risk in Adrenal Incidentalomas: Analysis of 2219 Patients. Ann Surg. 2022 Jan 1;275(1):e238-e244. doi: 10.1097/SLA.0000000000004048. PMID 32541223
- [Background] Balla A, Corallino D, Ortenzi M, Palmieri L, Meoli F, Guerrieri M, Paganini AM. Cancer risk in adrenalectomy: are adrenal lesions equal or more than 4 cm a contraindication for laparoscopy? Surg Endosc. 2022 Feb;36(2):1131-1142. doi: 10.1007/s00464-021-08380-7. Epub 2021 Mar 1. PMID 33650006
- [Background] Castillo OA, Vitagliano G, Secin FP, Kerkebe M, Arellano L. Laparoscopic adrenalectomy for adrenal masses: does size matter? Urology. 2008 Jun;71(6):1138-41. doi: 10.1016/j.urology.2007.12.019. Epub 2008 Mar 12. PMID 18336879
- See also: SICE website — https://siceitalia.com/
- Available data/document: Study Protocol: sice — https://siceitalia.com/ — SICE- Team di ricerca Endocrino-metabolica- crisal